CLINICAL TRIAL: NCT04156763
Title: A Comparison of Prism Cover Testing and a Virtual Reality Headset-based Test in the Objective Assessment of Ocular Deviation
Brief Title: Virtual Reality Test of Strabismus
Status: Terminated | Type: Observational
Why Stopped: CI has left the trust
Sponsor: Julie Dawson (Other)
Responsible Party: Sponsor-Investigator, Julie Dawson, Research Services Manager, Norfolk and Norwich University Hospitals NHS Foundation Trust
Organization: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Other Study IDs: 268329 (100-06-19)
Record Dates: First submitted 2019-11-06; First posted 2019-11-07 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Strabismus
Keywords: Strabismus Virtual Reality Prism Cover Test
MeSH Terms: conditions — Strabismus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Strabismus, or squint, describes any misalignment of the eyes, and can affect both children and adults. As a result, the images of the outside world conveyed to the brain from the two eyes do not correspond, which can result in diplopia, or 'double vision'. As well as impacting on a patient's functionality, strabismus can have cosmetic and psychosocial ramifications. Furthermore, if left untreated in childhood, strabismus can lead to life-long visual impairment, despite best spectacle correction.

Current treatment is guided by the exact nature of the strabismus and the patient's age; options include spectacle prescription to correct underlying refractive error, use of prisms to control deviation, or in certain cases, surgery. In order to investigate the size and type of strabismus present, and determine the best management, tests of ocular deviation are performed in Eye Clinics.

Quantitative objective assessment of the angle of horizontal and vertical strabismus is currently performed using the prism cover test - the patient is asked to look at a fixation target, and prisms of increasing power are placed in front of one eye until the ocular deviation is neutralised (i.e. there is no movement of the eyes to take up fixation). The test can provide accurate numerical recordings to aid in monitoring and surgical planning.

However, the prism cover test requires a range of different prisms, the presence of a near and distance fixation target, a trained examiner, and a patient able to fixate at an appropriate target without moving their head for the duration of the test. In this study, it will be investigated whether a virtual reality headset-based test can produce comparable measurements of ocular deviation to the traditional prism cover test, without the need for prisms, or control of head posture.

DETAILED DESCRIPTION:
Purpose

1. To establish whether a virtual reality headset-based test can produce accurate and reliable data on ocular deviation in those with disturbances of ocular motility, by comparing its performance to those of established tests of ocular deviation currently in use in clinical practice (prism cover test).
2. To assess the practicality, and subjective experience of a virtual reality headset- based Lancaster red-green test, using questionnaire surveys

Background

Strabismus, or squint, describes any misalignment of the eyes, and can affect both children and adults. As a result, the images of the outside world conveyed to the brain from the two eyes do not correspond, which can result in diplopia, or 'double vision'. As well as impacting on a patient's functionality, strabismus can have cosmetic and psychosocial ramifications. Furthermore, if left untreated in childhood, strabismus can lead to life-long visual impairment, despite best spectacle correction.

Current treatment is guided by the exact nature of the strabismus and the patient's age; options include spectacle prescription to correct underlying refractive error, use of prisms to control deviation, or in certain cases, surgery. In order to investigate the size and type of strabismus present, and determine the best management, tests of ocular deviation are performed in Eye Clinics.

Quantitative objective assessment of the angle of horizontal and vertical strabismus is currently performed using the prism cover test - the patient is asked to look at a fixation target, and prisms of increasing power are placed in front of one eye until the ocular deviation is neutralised (i.e. there is no movement of the eyes to take up fixation). The test can provide accurate numerical recordings to aid in monitoring and surgical planning.

However, the prism cover test requires a range of different prisms, the presence of a near and distance fixation target, a trained examiner, and a patient able to fixate at an appropriate target without moving their head for the duration of the test. In this study, it will be investigated whether a virtual reality headset-based test can produce comparable measurements of ocular deviation to the traditional prism cover test, without the need for prisms, or control of head posture.

Design and Methodology

Research participants will be recruited from the pool of patients presenting to the Eye department for their regular appointment.

Those who meet the inclusion criteria will have the study explained to them by a member of the research team in the department, and given a leaflet to read about the study. Should they wish to take part, they will have verbal and written consent taken, and then undergo two tests:

1. Prism cover test
2. Virtual reality headset-based test

Each test will last approximately 10 minutes. At the end of the two tests, they will be asked to fill in a questionnaire on their experience of the tests. They will require no additional visits to clinic as part of enrolling in the study.

Statistical Analysis

The angles of deviation of the eyes will be extracted from each of the three tests, and Bland Altman analysis will be applied to the data to check for agreement.

The subjective experience of the virtual reality headset-based Lancaster red-green test measured by the questionnaire, and compared to the subjective experience of the two established tests of ocular deviation using a paired t-test.

ELIGIBILITY:
Inclusion criteria:

• Patients with restrictive and paretic disturbances of ocular motility

Exclusion criteria:

* Patients without capacity to consent
* Patients unwilling to participate
* Patients aged under 18

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Research participants will be recruited from the pool of patients presenting to the Eye department for their regular appointment.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
The degree of agreement between the prism cover test and virtual reality headset-based test of ocular misalignment | 2 years
  The degree of agreement between the prism cover test and virtual reality headset-based test of ocular misalignment

SECONDARY OUTCOMES:
The subjective experience of the virtual reality headset-based test measured by questionnaire | 2 years
  The subjective experience of the virtual reality headset-based test measured by questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Norfolk & Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk, United Kingdom